CLINICAL TRIAL: NCT00127153
Title: A Comparative Study in Healthy Adults of the Safety, Tolerability, and Immunogenicity of V110 Formulated With Either All New Process Polysaccharides or All Current Process Polysaccharides
Brief Title: A Study of V110 a Pneumococcal Vaccine in Healthy Adults (V110-013)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: V110-013; 2005_039
Record Dates: First submitted 2005-08-02; First posted 2005-08-05 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Healthy; Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections | interventions — 2,4,5,4'-tetrachlorodiphenylsulfoxide; Pneumococcal Vaccines

INTERVENTIONS:
Biological: V110, pneumococcal vaccine polyvalent

SUMMARY:
The purpose of this trial is to evaluate the safety, tolerability, and immunogenicity of an investigational pneumococcal vaccine in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Males and females in good health, ages 20-40, with no history of pneumococcal vaccination

Exclusion Criteria:

* Subjects with a recent febrile illness
* Known or suspected immune dysfunction, conditions associated with immunosuppression, and receipt of immunosuppressive chemotherapy, including long-term corticosteroid therapy

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130
Dates: Start 2005-03; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Immunogenicity

SECONDARY OUTCOMES:
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC